CLINICAL TRIAL: NCT01216449
Title: Pharmacodynamics of Intravenous Citalopram in the Elderly: a Functional Magnetic Resonance Imaging Analysis
Brief Title: Effects of Intravenous (IV) Citalopram on Emotional Brain Activity in Healthy Young and Elderly Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: loss of funding
Sponsor: Rotman Research Institute at Baycrest (Other)
Collaborators: Centre for Addiction and Mental Health (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Bruce Pollock, VP Research, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 08-39
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Healthy Young and Elderly Volunteers
Keywords: Citalopram; Functional Magnetic Resonance Imaging; fMRI; Pharmacokinetics; Pharmacodynamics; Amygdala; Elderly
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Citalopram (Experimental)
  Interventions: Drug: Intravenous Citalopram
- Normal Saline (Placebo Comparator): 250mL of 0.9% Sodium Chloride Solution
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Intravenous Citalopram — Single dose of 20mg parenteral citalopram diluted in 250mL of 0.9% sodium chloride solution, infused over 30 minutes
  Arms: Intravenous Citalopram
Drug: Normal Saline — Single dose of 250mL of 0.9% sodium chloride solution, infused over 30 minutes
  Arms: Normal Saline

SUMMARY:
Antidepressant medications known as selective serotonin reuptake inhibitors (SSRIs) are most commonly prescribed to treat depression and anxiety. How antidepressants work on the brain to alter mood and behaviour is not well understood. This study will use a brain scanning technique (functional magnetic resonance imaging) to examine how aging impacts brain activation during emotional tasks after the administration of intravenous (IV) citalopram (this is the only SSRI available in this form, and is well tolerated and safe in young and old adults). The investigators will further determine what role genetic differences play in this relationship. The investigators expect to see an increase in brain signal as the concentration of IV citalopram increases. However, the investigators propose that the brain signal in older adults will not be as strong as in younger adults. Furthermore, the investigators expect that participants genetically predisposed to have fewer serotonin transporters (the site of action of SSRIs) will show greater decreases in brain activation with citalopram.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 60 or older (elderly group)
* Male aged 20-40 (younger adult group)
* English speaking
* Right-handed
* Non-smoker
* Score of 27 or greater on the Mini Mental State Exam

Exclusion Criteria:

* Unstable medical, cardiac, or neurological illness (including stroke, brain tumour, epilepsy, significant head injury, Alzheimer's, Parkinson's or Huntington's disease)
* Laboratory results indicating unanticipated illness or intolerability of blood drawing procedures or of study drug
* Current or lifetime Axis-I psychiatric diagnosis on the DSM-IV/SCID (i.e., Module A: Mood, Module F: Anxiety, Module B & C: Psychosis)
* History of drug or alcohol abuse within one year, or lifetime history of alcohol or drug dependence (i.e., SCID Module E: Substance Abuse, or clinically significant urine toxicology screen)
* History of non-tolerance to SSRI therapy; including history of SSRI-related syndrome of inappropriate antidiuretic hormone secretion (SIADH) or sinus bradycardia on ECG (less than 50 beats per minute)
* Contraindication to MRI (as per MRI Contraindication Screening Form)

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
BOLD fMRI Response | Visit 1, Visit 2
  Changes in affect-related neuronal activation as measured by blood oxygenation level-dependent (BOLD) fMRI response to IV citalopram are the primary outcome measures. Imaging data will be compared between IV citalopram and placebo administration and young and old adults.

SECONDARY OUTCOMES:
Genetics and Cognitive/Emotional Change | Visit 1, Visit 2
  Secondary measures include analysis of the relationship between 5HTT polymorphism and neuronal activation, and changes in cognitive and emotional assessments between IV citalopram and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G Pollock, MD PhD FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Rotman Research Institute at Baycrest, Toronto, Ontario, Canada